CLINICAL TRIAL: NCT02420743
Title: Third Trimester Serum Ferritin Concentration and Fetal MCA Peak Systolic Velocity as Predictors for Preterm Delivery
Brief Title: Serum Ferritin Concentration and Fetal MCA Doppler as Predictors for Preterm Delivery
Acronym: SFMCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Nesreen Abdel Fattah Abdullah Shehata, Lecturer of Obstetrics and Gynecology, Beni-Suef University
Other Study IDs: Beni-Suef 10
Record Dates: First submitted 2015-04-11; First posted 2015-04-20 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Preterm Delivery
Keywords: PTD
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: serum ferritin — serum ferritin will be measured serially at 26, 30 and 34 weeks gestation.
Procedure: MCA Doppler — MCA peak systolic value will be assessed at 26, 30 and 34 weeks gestation.

SUMMARY:
Pregnant women with iron deficiency anemia during third trimester will be assessed for serum ferritin and peak systolic value for fetal middle cerebral artery to find out their correlation with preterm delivery.

DETAILED DESCRIPTION:
Preterm delivery, defined as delivery before 37 weeks of completed gestation (259 days), is a major cause of neonatal morbidity and mortality. Despite extensive research, preterm birth still accounts for 5-10% of all deliveries in developed countries and rates are on the increase, including in the UK. While mortality associated with preterm delivery has declined due to use of antenatal steroids and improvements in neonatal intensive care, preterm babies still remain at risk of major complications. These include respiratory distress syndrome, necrotising enterocolitis, retinopathy of prematurity, sepsis, intraventricular haemorrhage, periventricular leucomalacia and long-term cognitive and sensory impairment. Two major determinants for the mortality and morbidity of babies born preterm are gestation at delivery and birthweight. Prematurity therefore carries significant cost implications to both healthcare services and society in general. High hemoglobin along with anemia was examined in an observational study. At entry to care, which ranged between 6 and 8.4 wk gestation, women with hemoglobin levels exceeding 130g/L had a greater than twofold increase in risk of preterm delivery and infant low birth weight. Neither risk was statistically significant, however, because of the small numbers with high hemoglobin. Similarly, a concentration of the iron storage protein, ferritin, that is high for the third trimester of pregnancy is also associated with an increased risk for preterm and very preterm delivery. Over the last twenty years, interest has been shown in using ultrasound parameters or Doppler studies of fetal blood to assess fetal anaemia. Middle cerebral artery Doppler has taken over and has replaced amniocentesis as a screening test for fetal anaemia in high risk pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant female from 24 weeks till 37 weeks gestation.
* Patients diagnosed as iron deficiency anemia.

Exclusion Criteria:

* Medical disorders as hypertension or diabetes.
* Kidney and liver diseases.
* Any other causes of anemia as haemoglobinopathies.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant females during third trimester. Women should be diagnosed as having iron deficiency anemia.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-10; Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
High serum ferritin concentration | at 26 to 34 weeks gestation
  The investigators will assess high serum ferritin concentration during third trimester and its effect on pregnancy outcome.

SECONDARY OUTCOMES:
PSV in fetal MCA doppler | 26 to 34 weeks gestation
  Peak systolic velocity of fetal MCA will be measured to diagnose fetal anemia and if correlated with preterm delivery.
Preterm delivery | From 34 to 37 weeks gestation
  The investigators will assess pregnancy outcome in the form og preterm delivery with abnormal parameters in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Nesreen A Shehata, MD, Study Director — Beni-Suef University
Locations (1):
- Nesreen Abdel Fattah Abdullah Shehata, Cairo, Fostat, Egypt

REFERENCES:
- [Background] Zhou LM, Yang WW, Hua JZ, Deng CQ, Tao X, Stoltzfus RJ. Relation of hemoglobin measured at different times in pregnancy to preterm birth and low birth weight in Shanghai, China. Am J Epidemiol. 1998 Nov 15;148(10):998-1006. doi: 10.1093/oxfordjournals.aje.a009577. PMID 9829872
- [Background] Mari G, Deter RL, Carpenter RL, Rahman F, Zimmerman R, Moise KJ Jr, Dorman KF, Ludomirsky A, Gonzalez R, Gomez R, Oz U, Detti L, Copel JA, Bahado-Singh R, Berry S, Martinez-Poyer J, Blackwell SC. Noninvasive diagnosis by Doppler ultrasonography of fetal anemia due to maternal red-cell alloimmunization. Collaborative Group for Doppler Assessment of the Blood Velocity in Anemic Fetuses. N Engl J Med. 2000 Jan 6;342(1):9-14. doi: 10.1056/NEJM200001063420102. PMID 10620643
- [Result] Stock SJ, Thomson AJ, Papworth S; Royal College of Obstetricians and Gynaecologists. Antenatal corticosteroids to reduce neonatal morbidity and mortality: Green-top Guideline No. 74. BJOG. 2022 Jul;129(8):e35-e60. doi: 10.1111/1471-0528.17027. Epub 2022 Feb 16. No abstract available. PMID 35172391
- [Result] Royal college of obstetricians and gynecologists. Preterm Prelabour Rupture of Membranes. Green-top Guideline No. 44. London: RCOG Press; 2010.